CLINICAL TRIAL: NCT00546910
Title: A Randomized, Double Blind Comparison of the Effects of Atomoxetine Versus Placebo on Neuropsychological Outcomes Across the Day in Children With Attention-Deficit/Hyperactivity Disorder (ADHD) by Use of a Computer Based Continuous Performance Test (cb CPT)
Brief Title: Comparison of Atomoxetine Versus Placebo in Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11148; B4Z-SB-LYDV (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): 0.5 milligram per kilogram (mg/kg) per day lead-in dose for 1 weeks followed by 7 weeks at 1.2 mg/kg per day dose.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Placebo matched to 1 week lead-in and 7 week standard target dose of atomoxetine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — A one-week atomoxetine treatment period with the 0.5 mg/kg per day lead-in dose will be succeeded by a 7 week period at the target dose of 1.2 mg/kg per day. 3 capsules of study medication have to be taken once daily in the morning, with or without food.
  Other Names: LY139603
  Arms: Atomoxetine
Drug: Placebo — 3 capsules of placebo have to be taken once daily in the morning, with or without food.
  Arms: Placebo

SUMMARY:
This is a two-arm, parallel, randomized, double-blind, placebo-controlled Phase 4 multicenter trial to compare the whole day efficacy of atomoxetine versus placebo in children aged 6 through 12 years with Attention-Deficit/Hyperactivity Disorder (ADHD) treated in an inpatient, day-patient and outpatient setting in Germany. Core symptoms will be measured during once or bi-weekly visits, three times per visit-day, by a computer based Continuous Performance Test. Following an initial 3-28-day screening and washout phase, patients will be assigned to double-blind treatment with atomoxetine or placebo. In the verum arm, a one-week atomoxetine treatment period with the 0.5 mg/kg per day lead-in dose will be succeeded by a 7 week period at the target dose of 1.2 mg/kg per day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are at least 6 years of age, and who will not have reached their 13th birthday
* Diagnosis of ADHD
* Normal intelligence
* Able to swallow capsules

Exclusion Criteria:

* Weight less than 20 kg or more than 60 kg at study entry
* Prior treatment with atomoxetine
* History of seizure disorder, suicidal risk, alcohol or drug abuse within the past 3 months
* History of severe allergies or multiple adverse drug reactions
* Cardiovascular disorders: hypertension, unexplained cardiac signs or symptoms, QT prolongation, inherited cardiac disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Germany (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Datteln
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dorsten
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eberswalde
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kehl
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolfenbüttel

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 63 | 62
Completed | 54 | 51
Not Completed | 9 | 11
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 5 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 63 | 62 | 125
Age Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.93) | 8.9 (1.64) | 9.0 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 47 | 50 | 97
Race/Ethnicity, Customized [Number; unit: participants] — Breakdown of participants by race
  participants
    Caucasian | 62 | 62 | 124
    African | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 63 | 62 | 125
Diagnosis [Number; unit: participants] — Breakdown of Attention Deficit/Hyperactivity Disorder (ADHD) diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
  participants
    ADHD-Combined Type | 40 | 48 | 88
    ADHD-Predominantly Inattentive Type | 17 | 11 | 28
    ADHD- Predominantly Hyperactive-Impulsive Type | 6 | 3 | 9
Number of Participants with Family History of ADHD [Number; unit: participants] — Number of participants with at least one biological relative (mother, father, sibling [brother, sister] or grandparent) with ADHD.
  participants
    At least one known relative with ADHD | 36 | 35 | 71
    None or missing | 27 | 27 | 54
Number of Participants with Prior Therapy For Attention-Deficit/Hyperactive Disorder (ADHD) [Number; unit: participants] — Summarizes number of participants who received previous medication and non-medication attention-deficit/hyperactive disorder (ADHD) therapy.
  participants
    Previous treatment for ADHD | 26 | 27 | 53
    None or missing | 37 | 35 | 72
Number of Participants with Psychiatric Comorbidities [Number; unit: participants] — Summarizes the psychologic comorbidities of participants. Because some participants may have one or more comorbidities while others may not, the breakdown of psychiatric comorbidities by treatment group does not equal the overall baseline number of participants in each treatment group.
  participants
    At least one psychiatric comorbidity | 25 | 25 | 50
    None or missing | 38 | 37 | 75
Summary Of Participants' Living Arrangements [Number; unit: participants] — Summarizes the participants' living arrangements according to where they live most of the time.
  participants
    Nuclear Family (Biological Mother and Father) | 38 | 36 | 74
    Single Mother | 15 | 17 | 32
    Step Parent (One Biologic and one step parent) | 10 | 9 | 19
ADHD Rating Scale-IV Parent Version: Investigator Administered & Scored, Total Score [Mean (Standard Deviation); unit: units on a scale] — ADHD Rating Scale-IV Parent Version: Investigator Administered & Scored (ADHD-RS-IV-PV:IR) measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
  units on a scale | 37.30 (10.62) | 36.68 (12.53) | 36.99 (11.56)
Clinical Global Impressions - Severity Of Attention Deficit Hyperactive Disorder Score [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions- Severity Of Attention Deficit Hyperactive Disorder (CGI-S-ADHD) measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
  units on a scale | 5.11 (1.02) | 5.05 (1.11) | 5.08 (1.06)
Time Since Initial Diagnosis Of ADHD [Mean (Standard Deviation); unit: years] | 1.8 (2.23) | 1.6 (1.89) | 1.7 (2.06)
Time Since Onset Of ADHD Symptoms [Mean (Standard Deviation); unit: years] | 4.9 (2.12) | 5.2 (1.95) | 5.0 (2.04)
Weekly Rating Of Evening & Morning Behavior-Revised-Investigator Rated, Total & Subscores [Mean (Standard Deviation); unit: units on a scale] — Weekly Rating Of Evening & Morning Behavior-Revised-Investigator Rated (WREMB-R-Inv) measures the level of difficulty of 11 common morning or evening behaviors (e.g. getting out of bed, doing homework, sitting through dinner). Possible scores for each item range from 0 (no difficulty) to 3 (a lot of difficulty) with a Total score (maximum score=33), Morning subscore (maximum score=9), Evening subscore (maximum score=24), and Item 11 score which pertains to degree of difficulty falling asleep (maximum score=3).
  units on a scale
    Total Score | 21.70 (7.64) | 21.58 (7.91) | 21.64 (7.75)
    Morning Subscore | 5.56 (2.66) | 4.63 (2.92) | 5.10 (2.82)
    Evening Subscore | 14.54 (4.76) | 15.39 (4.74) | 14.96 (4.75)
    Item 11 Subscore | 1.60 (1.23) | 1.56 (1.26) | 1.58 (1.24)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Computer-based Continuous Performance Test (cb- CPT; Qbtech AB, Sweden), Variable: Hyperactivity (Includes Time Active [TA], Distance [DIS], Area [AR], Microevents [ME], Motion Simplicity [MS]) Q-scores At Week 8
Description: Infra-red camera tracks movement of head reflector on patient performing computer test. Hyperactivity test variables: TA=percent time patient moved>1 centimeter (cm)/second; DIS=path of movement (m); AR=total area (cm2) of movements; ME=number of position changes>1 mm; MS=degree (percent) of directional changes. Results are converted to Q-scores (age and sex-adjusted normalized scores with a mean=0 and standard deviation (SD)=1 in general population, expressing the probability determined by the Gamma function in terms of SD of Gaussian density). Higher scores reflect more severe symptoms.
Time Frame: Baseline, 8 weeks (W8)
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Q-scores
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
Q-scores
  Baseline: TA-Morning | 0.62 (1.27) | 0.84 (0.84)
  Baseline: TA- Noon | 0.65 (1.13) | 0.76 (0.79)
  Baseline: TA- Evening | 0.66 (1.26) | 0.85 (0.83)
  W8 Change: TA- Morning | -0.32 (1.00) | 0.06 (0.84)
  W8 Change: TA- Noon | -0.60 (1.13) | 0.15 (0.74)
  W8 Change: TA- Evening | -0.55 (1.08) | 0.03 (0.76)
  Baseline: DIS- Morning | 1.41 (1.69) | 1.62 (1.68)
  Baseline: DIS- Noon | 1.55 (1.86) | 1.62 (1.74)
  Baseline: DIS- Evening | 1.47 (1.86) | 1.75 (1.73)
  W8 Change: DIS- Morning | -0.51 (1.80) | 0.38 (1.75)
  W8 Change: DIS- Noon | -1.06 (1.94) | 0.49 (1.52)
  W8 Change: DIS- Evening | -0.87 (1.71) | 0.07 (1.54)
  Baseline: AR- Morning | 1.14 (1.65) | 1.40 (1.56)
  Baseline: AR- Noon | 1.25 (1.66) | 1.45 (1.59)
  Baseline: AR- Evening | 1.19 (1.81) | 1.58 (1.67)
  W8 Change: AR- Morning | -0.38 (1.58) | 0.39 (1.60)
  W8 Change: AR- Noon | -0.87 (1.70) | 0.40 (1.18)
  W8 Change: AR- Evening | -0.71 (1.53) | -0.00 (1.45)
  Baseline: ME- Morning | 0.97 (1.32) | 1.15 (1.11)
  Baseline: ME- Noon | 0.98 (1.29) | 1.09 (1.19)
  Baseline: ME- Evening | 0.94 (1.45) | 1.18 (1.18)
  W8 Change: ME- Morning | -0.47 (1.42) | 0.20 (1.19)
  W8 Change: ME- Noon | -0.82 (1.48) | 0.28 (1.01)
  W8 Change: ME- Evening | -0.72 (1.41) | 0.06 (1.06)
  Baseline: MS- Morning | 0.21 (1.08) | 0.38 (1.01)
  Baseline: MS- Noon | 0.25 (1.12) | 0.32 (0.95)
  Baseline: MS- Evening | 0.22 (1.21) | 0.35 (1.05)
  W8 Change: MS- Morning | -0.22 (1.29) | -0.04 (1.07)
  W8 Change: MS- Noon | -0.39 (1.37) | -0.12 (0.94)
  W8 Change: MS- Evening | -0.38 (1.31) | -0.19 (1.09)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Time Active overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Time Active was tested at rank 8; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.52 to 0.87]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Distance overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Distance was tested at rank 5; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 1.27, 95% CI 2-sided [0.98 to 1.57]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Area overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Area was tested at rank 6; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.81 to 1.35]
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Microevents overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Microevents was tested at rank 3; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [0.78 to 1.22]
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Motion Simplicity overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Motion Simplicity was tested at rank 9; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.18 to 0.58]

2. Secondary Outcome: Change From Baseline Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator-Administered And Scored (ADHDRS-IV-Parent:Inv) Total Score At Week 8
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
Time Frame: Baseline, 8 weeks
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
units on a scale
  Baseline to Visit 7 (Week 8) | -17.19 (15.63) | -4.76 (11.51)
  Baseline to LOCF | -15.78 (15.19) | -4.21 (10.89)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Comparison of atomoxetine vs. placebo at Visit 7 (Week 8); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for ADHD-RS Total Score; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 11.60, 95% CI 2-sided [8.20 to 14.99]

3. Secondary Outcome: Change From Baseline Clinical Global Impressions-Severity of ADHD (CGI-S-ADHD) Score at Week 8
Description: CGI-S-ADHD measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline, 8 weeks
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
units on a scale
  Baseline to Visit 7 (Week 8) | -1.78 (1.61) | -0.63 (1.11)
  Baseline to LOCF | -1.52 (1.63) | -0.40 (1.17)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Comparison of atomoxetine vs. placebo at Visit 7 (Week 8); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for CGI-S ADHD score; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [0.76 to 1.46]

4. Secondary Outcome: Change From Baseline Weekly Rating Of Evening and Morning Behavior-Revised-Investigator Rated, Total and Subscores at Week 8
Description: Weekly Rating Of Evening & Morning Behavior-Revised-Investigator Rated (WREMB-R-Inv) measures the level of difficulty of 11 common morning or evening behaviors (e.g. getting out of bed, doing homework, sitting through dinner). Possible scores for each item range from 0 (no difficulty) to 3 (a lot of difficulty) with a Total score (maximum score=33), Morning subscore (maximum score=9), Evening subscore (maximum score=24), and Item 11 score which pertains to degree of difficulty falling asleep (maximum score=3).
Time Frame: Baseline, 8 weeks
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
units on a scale
  Total Score: Baseline to Visit 7 (Week 8) | -10.72 (10.21) | -5.10 (6.83)
  Total Score: Baseline to LOCF | -9.59 (9.98) | -3.90 (7.83)
  Evening Subscore: Baseline to Visit 7 (Week 8) | -6.91 (6.38) | -3.57 (4.36)
  Evening Subscore: Baseline to LOCF | -6.30 (6.21) | -3.03 (5.18)
  Morning Subscore: Baseline to Visit 7 (Week 8) | -2.81 (3.04) | -1.16 (2.74)
  Morning Subscore: Baseline to LOCF | -2.46 (3.00) | -0.65 (2.94)
  Item 11 Subscore: Baseline to Visit 7 (Week 8) | -1.00 (1.60) | -0.37 (1.00)
  Item 11 Subscore: Baseline to LOCF | -0.83 (1.60) | -0.23 (1.05)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Total Score; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 5.74, 95% CI 2-sided [3.55 to 7.92]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — P-value for Evening subscore; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 3.96, 95% CI 2-sided [2.49 to 5.44]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.002, Mixed Models Analysis — P-value for Morning subscore; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [0.42 to 1.93]
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Item 11 (difficulty falling asleep); Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [0.31 to 0.93]

5. Primary Outcome: Change From Baseline cb CPT Variable: Inattention (Includes Reaction Time Variation[RTV], Omission Error [OR], Mean Reaction Time [mRT], Normalized Variation Of Reaction Time [nVRT]) Q-scores At Week 8
Description: Computer test. Patient is to press button if target appears, but not at non-target. Inattention test variables: mRT=average time (ms) from target presentation to response; RTV=standard deviation of mRT; nVRT=RTV expressed in terms of RT (variation as a percent of mean value); OE= percent of omitted targets. Results are converted to Q-scores (age and sex-adjusted normalized scores with a mean=0 and SD=1 in the general population, expressing the probability determined by the Gamma function in terms of SD of Gaussian density). Higher scores reflect more severe symptoms.
Time Frame: Baseline, 8 weeks
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Q-scores
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
Q-scores
  Baseline: RTV-Morning | 2.93 (2.41) | 2.49 (1.62)
  Baseline: RTV-Noon | 2.95 (2.11) | 2.48 (1.92)
  Baseline: RTV-Evening | 2.63 (2.49) | 2.19 (2.00)
  W8: RTV-Morning | -0.89 (2.29) | -0.09 (1.78)
  W8: RTV-Noon | -1.07 (1.92) | 0.00 (1.70)
  W8: RTV-Evening | -0.90 (1.98) | -0.00 (1.88)
  Baseline: OR- Morning | 1.12 (1.24) | 1.13 (1.19)
  Baseline: OR- Noon | 1.31 (1.32) | 1.30 (1.32)
  Baseline: OR- Evening | 1.22 (1.43) | 1.28 (1.34)
  W8: OR- Morning | 0.01 (1.83) | 0.54 (1.14)
  W8: OR- Noon | 0.03 (1.45) | 0.53 (1.17)
  W8: OR- Evening | -0.04 (1.50) | 0.52 (1.20)
  Baseline: mRT- Morning | 2.42 (2.03) | 1.92 (1.53)
  Baseline: mRT- Noon | 2.40 (1.78) | 2.02 (1.49)
  Baseline: mRT- Evening | 2.23 (1.77) | 1.86 (1.49)
  W8: mRT- Morning | -0.18 (1.84) | 0.35 (1.28)
  W8: mRT- Noon | -0.35 (1.53) | 0.12 (1.42)
  W8: mRT- Evening | -0.13 (1.40) | 0.48 (1.37)
  Baseline: nVRT-Morning | 1.00 (1.60) | 0.93 (1.28)
  Baseline: nVRT-Noon | 1.06 (1.48) | 0.82 (1.26)
  Baseline: nVRT-Evening | 0.92 (1.81) | 0.68 (1.31)
  W8: nVRT-Morning | -0.59 (1.58) | -0.36 (1.15)
  W8: nVRT-Noon | -0.65 (1.48) | -0.09 (0.97)
  W8: nVRT-Evening | -0.65 (1.75) | -0.33 (1.19)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Reaction Time Variation overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Reaction time variation was tested at rank 1; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [0.66 to 1.35]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Omission Error overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Omission error was tested at rank 7; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [0.46 to 0.93]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Mean Reaction Time overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Mean reaction time was tested at rank 2; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.17 to 0.65]
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Normalized Variation of Reaction Time overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Normalized Variation of Reaction Time was tested at rank 10; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [0.26 to 0.73]

6. Primary Outcome: Change From Baseline cb CPT Variable: Impulsivity (Includes Commission Error [CE], Anticipatory Response [AR]) Q-scores At Week 8
Description: Computer test. Patient is to press button if target appears, but not at non-target. Impulsivity variables during test: CE=percent of response to non-target; ANT=percent of responses prior to target presentation. Results are converted to Q-scores (age and sex-adjusted normalized scores with a mean=0 and standard deviation=1 in the general population, expressing the probability determined by the Gamma function in terms of standard deviation of Gaussian density). Higher scores reflect more severe symptoms.
Time Frame: Baseline, 8 weeks
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Q-scores
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
Q-scores
  Baseline: CE- Morning | -0.68 (1.34) | -0.89 (1.03)
  Baseline: CE- Noon | -0.65 (1.29) | -0.85 (0.94)
  Baseline: CE- Evening | -0.80 (1.23) | -0.87 (1.06)
  W8: CE- Morning | -0.88 (1.33) | -0.32 (0.90)
  W8: CE- Noon | -0.94 (1.33) | -0.44 (0.82)
  W8: CE- Evening | -0.76 (1.31) | -0.49 (0.92)
  Baseline: AR- Morning | 0.41 (1.15) | 0.15 (0.88)
  Baseline: AR- Noon | 0.28 (1.06) | 0.12 (0.85)
  Baseline: AR- Evening | 0.32 (1.16) | 0.08 (0.85)
  W8: AR- Morning | -0.50 (0.98) | -0.34 (0.84)
  W8: AR-Noon | -0.54 (0.87) | -0.31 (0.84)
  W8: AR- Evening | -0.52 (0.83) | -0.28 (0.78)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Commission Error overall for morning, noon and evening. Primary tests were performed hierarchically to adjust for multiplicity. Commission Error was tested at rank 4; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [0.31 to 0.68]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — P-value is for Anticipatory Response overall for morning, noon and evening. Anticipatory Response was not tested in the primary analysis but is a secondary endpoint; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.02 to 0.31]

7. Primary Outcome: Change From Baseline cb CPT Variable: Other (Includes Error Rate [ER] and Multi Response [MR]) Q-scores At Week 8
Description: Computer test. Patient is to press button if target appears, but not at non-target. Other variables during test: ER=percent of overall incorrect responses (CE and OE); MR=percent of multiple responses per presentation of target (patient responds more than once to target). Results are converted to Q-scores (age and sex-adjusted normalized scores with a mean=0 and standard deviation=1 in the general population, expressing the probability determined by the Gamma function in terms of standard deviation of Gaussian density). Higher scores reflect more severe symptoms.
Time Frame: Baseline, 8 weeks
Population: Full analysis population (N=125) including all randomized participants taking at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Q-scores
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 63 | 62
Q-scores
  Baseline: ER- Morning | 0.37 (1.56) | 0.30 (1.15)
  Baseline: ER- Noon | 0.52 (1.46) | 0.41 (1.24)
  Baseline: ER- Evening | 0.37 (1.58) | 0.41 (1.24)
  W8: ER- Morning | -0.41 (2.06) | 0.35 (1.10)
  W8: ER- Noon | -0.44 (1.70) | 0.32 (1.06)
  W8: ER- Evening | -0.43 (1.80) | 0.28 (1.10)
  Baseline: MR- Morning | -0.04 (1.25) | -0.26 (0.84)
  Baseline: MR- Noon | 0.01 (1.15) | -0.30 (0.95)
  Baseline: MR- Evening | 0.03 (1.25) | -0.34 (0.89)
  W8: MR- Morning | -0.23 (1.15) | -0.24 (0.78)
  W8: MR- Noon | -0.45 (0.97) | -0.16 (0.83)
  W8: MR- Evening | -0.35 (1.30) | -0.16 (0.77)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for Error Rate overall for morning, noon and evening. Error Rate was not tested in the primary analysis but is a secondary endpoint; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.69 to 1.18]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.178, Mixed Models Analysis — P-value is for Multi Response overall for morning, noon and evening. Multi Response was not tested in the primary analysis but is a secondary endpoint; Positive values for the mean difference are in favor of the atomoxetine arm; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.05 to 0.28]

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 32/63 | 27/62
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=63) | Placebo (N=62)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 4 (4) | 1 (2)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Aggression (Psychiatric disorders) | 0 (0) | 4 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days